CLINICAL TRIAL: NCT00924053
Title: A Phase I, Randomized, Placebo-Controlled Study to Assess the Safety, Tolerability and Pharmacokinetics of EGT0001474 in Subjects With Type 2 Diabetes
Brief Title: Safety, Tolerability and Pharmacokinetics Study of EGT0001474 in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Theracos (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: THR-1474-C-396
Record Dates: First submitted 2009-06-16; First posted 2009-06-18 (Estimated); Results first posted 2011-08-17 (Estimated); Last update posted 2019-06-17 (Actual); Status verified 2019-06

CONDITIONS: Diabetes Mellitus Type 2
Keywords: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EGT0001474 (Experimental)
  Interventions: Drug: EGT0001474
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EGT0001474 — Cohort 1: single dose of 25 mg EGT0001474 given as an oral capsule; Cohort 2: single dose of 75 mg EGT0001474 given as 3 oral capsules; Cohort 3: single dose of 150 mg EGT0001474 given as 6 oral capsules.
  Other Names: Human SGLT2 inhibitor
  Arms: EGT0001474
Drug: Placebo — Placebo capsules to match EGT0001474
  Other Names: Human SGLT2 inhibitor
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the safety, tolerability and pharmacokinetics (how much of the drug gets into the blood and how long it takes the body to get rid of it) of single doses of EGT0001474 given to patients with Type 2 diabetes. The study will also evaluate how EGT0001474 affects the amount of glucose produced by the body in the urine.

DETAILED DESCRIPTION:
EGT0001474 is a compound that may inhibit the effect of other compounds in the body known as sugar transporters. The use of EGT0001474 may enhance the elimination of glucose from the blood by increasing the amount of urine produced. This would help prevent an abnormal decrease in blood sugar (hypoglycemia) both during fasting and after meals without increasing insulin secretion (which may result in weight gain or an abnormal increase in blood sugar known as Type 2 diabetes).

ELIGIBILITY:
Inclusion Criteria:

* Male or females between the ages of 18 to 70 diagnosed with Type 2 diabetes.
* Body mass Index (BMI) between 18 kg/m2 and 37 kg/m2.
* HbA1c levels between 6.5 and 9.0 (inclusive) where the upper limit of normal for the HbA1c assay is 6.4% or 6.2-9.0% (inclusive) where the upper limit of normal for the HbA1c assay is 6.1% and fasting plasma glucose between 110 and 240 mg/dL (inclusive) while on diabetic medications.
* If taking drugs for diabetes, must be medically able and willing to discontinue diabetes medications for the duration of the study.
* Female subjects must be surgically sterilized or postmenopausal.
* Non-smoker for at least 3 months.
* Negative alcohol screen.

Exclusion Criteria:

* Type 1 diabetes.
* Use of insulin therapy or oral antidiabetic medication other than metformin, sitagliptin or a sulfonylurea.
* Sitting blood pressure above 150/95 mmHg on 2 evaluations at least 10 minutes apart at screening.
* Treatment with an investigational drug within 30 days or 7 half-lives, whichever is longer.
* Previous treatment with EGT0001474.
* Vaccination within 30 days prior to the first dose of study medication.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-06; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mason W. Freeman, M.D., Study Chair — Massachusetts General Hospital
Locations (1):
- dgd Research Inc., a Cetero Research Company, San Antonio, Texas, United States

REFERENCES:
- [Background] Blondel O, Bailbe D, Portha B. Insulin resistance in rats with non-insulin-dependent diabetes induced by neonatal (5 days) streptozotocin: evidence for reversal following phlorizin treatment. Metabolism. 1990 Aug;39(8):787-93. doi: 10.1016/0026-0495(90)90120-2. PMID 2198430
- [Background] Cowie CC, Rust KF, Byrd-Holt DD, Eberhardt MS, Flegal KM, Engelgau MM, Saydah SH, Williams DE, Geiss LS, Gregg EW. Prevalence of diabetes and impaired fasting glucose in adults in the U.S. population: National Health And Nutrition Examination Survey 1999-2002. Diabetes Care. 2006 Jun;29(6):1263-8. doi: 10.2337/dc06-0062. PMID 16732006
- [Background] American Diabetes Association. Economic costs of diabetes in the U.S. In 2007. Diabetes Care. 2008 Mar;31(3):596-615. doi: 10.2337/dc08-9017. PMID 18308683
- [Background] American Diabetes Association. Standards of medical care in diabetes--2008. Diabetes Care. 2008 Jan;31 Suppl 1:S12-54. doi: 10.2337/dc08-S012. No abstract available. PMID 18165335
- [Background] Ehrenkranz JR, Lewis NG, Kahn CR, Roth J. Phlorizin: a review. Diabetes Metab Res Rev. 2005 Jan-Feb;21(1):31-8. doi: 10.1002/dmrr.532. PMID 15624123
- [Background] Han S, Hagan DL, Taylor JR, Xin L, Meng W, Biller SA, Wetterau JR, Washburn WN, Whaley JM. Dapagliflozin, a selective SGLT2 inhibitor, improves glucose homeostasis in normal and diabetic rats. Diabetes. 2008 Jun;57(6):1723-9. doi: 10.2337/db07-1472. Epub 2008 Mar 20. PMID 18356408
- [Background] Jabbour SA, Goldstein BJ. Sodium glucose co-transporter 2 inhibitors: blocking renal tubular reabsorption of glucose to improve glycaemic control in patients with diabetes. Int J Clin Pract. 2008 Aug;62(8):1279-84. doi: 10.1111/j.1742-1241.2008.01829.x. PMID 18705823
- [Background] Komoroski B, Vachharajani N, Feng Y, Li L, Kornhauser D, Pfister M. Dapagliflozin, a novel, selective SGLT2 inhibitor, improved glycemic control over 2 weeks in patients with type 2 diabetes mellitus. Clin Pharmacol Ther. 2009 May;85(5):513-9. doi: 10.1038/clpt.2008.250. Epub 2009 Jan 7. PMID 19129749
- [Background] Krook A, Kawano Y, Song XM, Efendic S, Roth RA, Wallberg-Henriksson H, Zierath JR. Improved glucose tolerance restores insulin-stimulated Akt kinase activity and glucose transport in skeletal muscle from diabetic Goto-Kakizaki rats. Diabetes. 1997 Dec;46(12):2110-4. doi: 10.2337/diab.46.12.2110. PMID 9392506
- [Background] Oku A, Ueta K, Arakawa K, Ishihara T, Nawano M, Kuronuma Y, Matsumoto M, Saito A, Tsujihara K, Anai M, Asano T, Kanai Y, Endou H. T-1095, an inhibitor of renal Na+-glucose cotransporters, may provide a novel approach to treating diabetes. Diabetes. 1999 Sep;48(9):1794-800. doi: 10.2337/diabetes.48.9.1794. PMID 10480610
- [Background] Pajor AM, Wright EM. Cloning and functional expression of a mammalian Na+/nucleoside cotransporter. A member of the SGLT family. J Biol Chem. 1992 Feb 25;267(6):3557-60. PMID 1740408
- [Background] Santer R, Kinner M, Lassen CL, Schneppenheim R, Eggert P, Bald M, Brodehl J, Daschner M, Ehrich JH, Kemper M, Li Volti S, Neuhaus T, Skovby F, Swift PG, Schaub J, Klaerke D. Molecular analysis of the SGLT2 gene in patients with renal glucosuria. J Am Soc Nephrol. 2003 Nov;14(11):2873-82. doi: 10.1097/01.asn.0000092790.89332.d2. PMID 14569097
- [Background] Toggenburger G, Kessler M, Semenza G. Phlorizin as a probe of the small-intestinal Na+,D-glucose cotransporter. A model. Biochim Biophys Acta. 1982 Jun 14;688(2):557-71. doi: 10.1016/0005-2736(82)90367-4. PMID 7201854
- [Background] Tsujihara K, Hongu M, Saito K, Inamasu M, Arakawa K, Oku A, Matsumoto M. Na(+)-glucose cotransporter inhibitors as antidiabetics. I. Synthesis and pharmacological properties of 4'-dehydroxyphlorizin derivatives based on a new concept. Chem Pharm Bull (Tokyo). 1996 Jun;44(6):1174-80. doi: 10.1248/cpb.44.1174. PMID 8814948

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first subject was enrolled on 12 Jun 2009; the last subject was completed on 28 Jul 2009. Subjects participated at a CRO in San Antonio, TX.
Pre-assignment Details: For 3 weeks after enrollment and prior to assignment to treatment and receiving drug, subjects were screened (informed consent, medical history, vital signs, electrocardiogram, laboratory test results, and screening for drugs of abuse and alcohol use) and began a 14 day washout period (counseling, review of medications and adverse events).
Groups:
- Placebo: Received 1, 3, or 6 placebo capsules once daily.
- EGT0001474 25 mg: Received one 25 mg capsule once daily.
- EGT0001474 75 mg: Received three 25mg capsules once daily.
- EGT0001474 150mg: Received six 25 mg capsules once daily.
Period: Overall Study
Arm/Group | Placebo | EGT0001474 25 mg | EGT0001474 75 mg | EGT0001474 150mg
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | EGT0001474 25 mg | EGT0001474 75 mg | EGT0001474 150mg | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 6 | 6 | 24
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 4 | 3 | 12
  Male | 4 | 3 | 2 | 3 | 12

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of EGT0001474
Description: Safety and tolerability were measured in terms of the number of mild, moderate and severe adverse events experienced by any participants.
Time Frame: 25 days
Population: All patients who took study medication were included in the analysis.
Measure: Number; unit: Events
Arm/Group | Placebo | EGT0001474 25 mg | EGT0001474 75 mg | EGT0001474 150mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
Events
  Mild adverse events | 5 | 0 | 9 | 3
  Moderate adverse events | 0 | 0 | 0 | 1
  Serious adverse events | 0 | 0 | 0 | 0

2. Primary Outcome: AUC 0-t
Description: Area under the plasma concentration-time curve from time 0 to time t
Time Frame: 3 days
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Placebo | EGT0001474 25 mg | EGT0001474 75 mg | EGT0001474 150mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
ng*hr/mL | NA (NA) — Placebo did not receive EGT0001474 drug | 1103.89 (470.31) | 3370.29 (499.36) | 6177.8 (1691.04)

3. Primary Outcome: AUC0-24
Description: Area under the plasma concentration-time curve from time 0 to hour 24
Time Frame: 3 days
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Placebo | EGT0001474 25 mg | EGT0001474 75 mg | EGT0001474 150mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
ng*hr/mL | NA (NA) — Placebo did not receive EGT0001474 drug | 987.3 (368.21) | 2990.63 (461.18) | 5584.72 (1516.64)

4. Primary Outcome: AUC Inf
Description: Area under the plasma concentration-time curve from time 0 to infinity
Time Frame: 3 days
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Placebo | EGT0001474 25 mg | EGT0001474 75 mg | EGT0001474 150mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
ng*hr/mL | NA (NA) — Placebo did not receive EGT0001474 drug | 1165.59 (479.88) | 3532.02 (524.74) | 6399.55 (1736.38)

5. Primary Outcome: Cmax
Description: Maximum plasma concentration
Time Frame: 3 days
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo | EGT0001474 25 mg | EGT0001474 75 mg | EGT0001474 150mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
ng/mL | NA (NA) — Placebo did not receive EGT0001474 drug | 157.23 (76.25) | 518.67 (176.36) | 1014 (372.63)

6. Primary Outcome: Tmax
Description: Time of maximum plasma concentration
Time Frame: 3 days
Measure: Median (Full Range); unit: hour
Arm/Group | Placebo | EGT0001474 25 mg | EGT0001474 75 mg | EGT0001474 150mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
hour | NA [NA to NA] — Placebo did not receive EGT0001474 drug | 3 [1 to 8] | 2 [1 to 6] | 2 [0.5 to 6]

7. Primary Outcome: λz
Description: Terminal phase rate constant
Time Frame: 3 days
Measure: Mean (Standard Deviation); unit: 1/hour
Arm/Group | Placebo | EGT0001474 25 mg | EGT0001474 75 mg | EGT0001474 150mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
1/hour | NA (NA) — Placebo did not receive EGT0001474 drug | 0.0741 (0.0215) | 0.0613 (0.0168) | 0.0622 (0.0195)

8. Primary Outcome: t1/2
Description: Apparent terminal half life
Time Frame: 3 days
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Placebo | EGT0001474 25 mg | EGT0001474 75 mg | EGT0001474 150mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
hour | NA (NA) — Placebo did not receive EGT0001474 drug | 10.1 (3.21) | 12.18 (3.88) | 12.15 (3.94)

9. Primary Outcome: CL/F
Description: The apparent rate of oral clearance of EGT0001474.Oral clearance was defined as rate of drug removal from the body after oral administration.
Time Frame: 3 days
Measure: Mean (Standard Deviation); unit: mL/hr
Arm/Group | Placebo | EGT0001474 25 mg | EGT0001474 75 mg | EGT0001474 150mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
mL/hr | NA (NA) — Placebo did not receive EGT0001474 drug | 24479.26 (9146.52) | 21616.42 (3112.38) | 24996.33 (7009.45)

10. Primary Outcome: Vz/F
Description: Apparent volume of distribution
Time Frame: 3 days
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Placebo | EGT0001474 25 mg | EGT0001474 75 mg | EGT0001474 150mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
mL | NA (NA) — Placebo did not receive EGT0001474 drug | 348376.12 (15666.55) | 382783.75 (138953.19) | 435944.78 (179821.44)

ADVERSE EVENTS:
Time Frame: 25 days total (14 day washout, 4 days in study, 1 week follow up after dosing)
Arm/Group | Placebo | EGT0001474 25 mg | EGT0001474 75 mg | EGT0001474 150mg
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 2/6 | 0/6 | 4/6 | 2/6
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo (N=6) | EGT0001474 25 mg (N=6) | EGT0001474 75 mg (N=6) | EGT0001474 150mg (N=6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood triglyceride increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 3 (4) | 2 (2)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0/0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Nervous system disorders) | 0/0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Vessel puncture site haematoma (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site reaction (General disorders) | 1 (1) | 0 (0) | 0/0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes